CLINICAL TRIAL: NCT03295396
Title: A Phase II, Open-label Study of ONC201 in Adults With Recurrent High-grade Glioma
Brief Title: ONC201 in Adults With Recurrent H3 K27M-mutant Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor terminated the study to prioritize enrollment in a randomized Phase 3 trial of ONC201 in an earlier setting. This decision was unrelated to any safety concerns with dordaviprone (ONC201).
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC013
Record Dates: First submitted 2017-08-01; First posted 2017-09-27 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patients received 625 mg dordaviprone (ONC201) once weekly.
  Arm A included patients with recurrent H3 K27M-mutant glioma including those with diffuse intrinsic pontine glioma (DIPG), primary spinal tumors, and some atypical histologies.
  Interventions: Drug: Dordaviprone (ONC201)
- Arm B (Experimental): Patients received 625 mg dordaviprone (ONC201) once weekly.
  Arm B included patients with recurrent H3 K27M-mutant glioma, but excluded patients with the following:
  * Primary malignant lesion located in the pons or spinal cord.
  * Atypical non-astrocytic histologies such as ependymoma, ganglioma and pleomorphic xanthoastrocytoma, or pilocytic astrocytoma and subependymal giant cell astrocytoma (SEGA).
  * Prior bevacizumab treatment of >4 doses of >7.5 mg/kg
  Interventions: Drug: Dordaviprone (ONC201)

INTERVENTIONS:
Drug: Dordaviprone (ONC201) — Dordaviprone (ONC201) is a central nervous system (CNS)-penetrant, small-molecule imipridone that acts as a mitochondrial caseinolytic protease P (ClpP) agonist and a dopamine receptor D2 (DRD2) antagonist.
  Other Names: Dordaviprone

SUMMARY:
This was a Phase 2, open-label, 2-arm study of dordaviprone (ONC201) in patients with recurrent H3 K27M- mutant glioma.

The primary assessment of dordaviprone (ONC201) involved evaluating its anti-tumor activity through the overall response rate according to the Response Assessment in Neuro-Oncology (RANO) criteria for high-grade glioma (HGG).

DETAILED DESCRIPTION:
This study included 2 arms:

* Arm A included patients with recurrent H3 K27M-mutant glioma.
* Arm B included patients with recurrent H3 K27M-mutant glioma, but excluded patients with the following:

  * Primary malignant lesion located in the pons or spinal cord.
  * Atypical non-astrocytic histologies such as ependymoma, ganglioma and pleomorphic xanthoastrocytoma, or pilocytic astrocytoma and subependymal giant cell astrocytoma (SEGA).
  * Prior bevacizumab treatment of >4 doses of >7.5 mg/kg

Patients received dordaviprone (ONC201) 625 mg once weekly.

The primary assessment of dordaviprone (ONC201) involved evaluating its anti-tumor activity through the overall response rate according to the Response Assessment in Neuro-Oncology (RANO) criteria for high-grade glioma (HGG). Safety was also assessed, with evaluations including the reporting of adverse events, as well as measurements of vital signs and clinical laboratory results.

This study was terminated by an administrative protocol amendment (17 January 2023). The decision to terminate the study was not related to any safety concerns with dordaviprone (ONC201). Before the study was terminated, a total of 73 patients were enrolled and received at least 1 dose of dordaviprone (ONC201).

ELIGIBILITY:
Inclusion Criteria:

1. Had histologically confirmed diagnosis of high-grade glioma (HGG) in any tumor sample and presence of histone H3 K27M mutation detected in a Clinical Laboratory Improvement Amendment (CLIA) certified laboratory by immunohistochemistry or DNA sequencing test on any glioma tumor sample.
2. Had unequivocal evidence of progressive disease on contrast-enhanced brain computed tomography (CT) or magnetic resonance imaging (MRI) as defined by Response Assessment in Neuro-Oncology (RANO)-HGG criteria, or have documented recurrent glioma on diagnostic biopsy.
3. Had measurable disease by RANO-HGG criteria.
4. Patients must have had previous therapy with at least radiotherapy.
5. Had no more than two prior episodes of recurrence from radiotherapy and/or chemotherapy. Use of bevacizumab solely for treatment of radiation necrosis, pseudoprogression, or treatment effect was not considered a recurrence.
6. Had an interval of at least 90 days from the completion of radiotherapy to the first dose of dordaviprone (ONC201). If patients were within 90 days of radiotherapy, they may have still been eligible if they met one or more of the following criteria.

   1. Progressive tumor is outside the original high-dose radiotherapy target volume as determined by the treating investigator, or
   2. Histologic confirmation of tumor through biopsy or resection, or
   3. Nuclear medicine imaging, magnetic resonance (MR) spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than pseudoprogression or radiation necrosis obtained within 28 days of registration.
7. From the projected start of scheduled study treatment, the following time periods must have had elapsed: 5 half-lives from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies.
8. All adverse events Grade >1 related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must have been resolved to Grade 1 or baseline, except for alopecia and sensory neuropathy Grade ≤2, or other Grade ≤2 not constituting a safety risk based on investigator's judgment, are acceptable.
9. Were male or female aged ≥18 years.
10. Had a Karnofsky Performance Status (KPS) ≥60.
11. Had adequate organ and marrow function as defined below, all screening labs should be performed within 14 days of treatment initiation:

    * leukocytes ≥ 3,000/mcL
    * absolute neutrophil count ≥ 1,500/mcL
    * platelets ≥ 75,000/mcL
    * hemoglobin > 8.0 mg/dL
    * total bilirubin ≤ 2.0 × upper limit of normal (ULN)
    * aspartate aminotransferase (AST) [SGOT]/alanine aminotransferase (ALT) [SGPT] ≤ 2.5 × ULN
    * creatinine ≤ULN OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above normal.
12. Had contrast-enhanced head CT or brain MRI and entire spine MRI within 14 days prior to start of study drug.
13. Corticosteroid dose must have been stable or decreasing for at least 3 days prior to the baseline CT or MRI scan.
14. Women of childbearing potential (WOCBP) and men must have agreed to use adequate contraception prior to study entry and for the duration of study participation and for 30 days after the last dose of therapy. Highly effective contraceptive measures include: stable use of oral contraceptives such as combined estrogen and progestogen and progestogen only hormonal contraception or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; intrauterine hormone-releasing system (IUS); bilateral tubal ligation; vasectomy and sexual abstinence.

    1. WOCBP must have had a negative serum or urine pregnancy test within 28 days of initiation of dosing.
    2. Contraception was not required for men with documented vasectomy.
    3. Postmenopausal women must have been amenorrheic for at least 12 months in order not to be considered of childbearing potential.
    4. Pregnancy testing and contraception were not required for women with documented hysterectomy or tubal ligation.
15. Had availability of a paraffin-embedded or frozen tumor-tissue block with a minimum of 1 cm2 of tumor surface area, or 20 unstained slides from the tumor tissue specimen if a tumor block cannot be submitted. If a patient has had only a stereotactic biopsy, then 5 unstained slides may be accepted with prior approval from the Sponsor, however all efforts must be made to obtain as close to 20 slides as possible.
16. Had the ability to be able to swallow and retain orally administered medication
17. Had the ability to understand and the willingness to sign a written informed consent document. Only patients who had capacity to consent were enrolled in the study.

Exclusion Criteria:

1. Arm B: Had a primary malignant lesion located in the pons or spinal cord.
2. Arm B: Had atypical non-astrocytic histologies such as ependymoma, ganglioma and pleomorphic xanthoastrocytoma, or pilocytic astrocytoma and subependymal giant cell astrocytoma (SEGA).
3. Arm B: Had prior bevacizumab treatment of >4 doses of >7.5 mg/kg
4. Had a history of allergic reactions attributed to compounds of similar chemical or biologic composition to dordaviprone (ONC201) or its excipients.
5. Had current or planned participation in a study of an investigational agent or using an investigational device.
6. Had presence of diffuse leptomeningeal disease or evidence of cerebrospinal fluid (CSF) dissemination.
7. Had uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
8. Had an active infection requiring systemic therapy.
9. Were pregnant and/or breastfeeding women or unable to maintain use of contraception while on study and for 30 days after the last dose of study drug. Dordaviprone (ONC201) is a novel agent with unknown potential for teratogenic or abortifacient effects.
10. Had known HIV-positive test on combination antiretroviral therapy.
11. Had known history of cardiac arrhythmias including atrial fibrillation, tachyarrhythmias or bradycardia, unless arrhythmia is controlled and after Cardiology has cleared patient to receive dordaviprone (ONC201). Receiving therapeutic agents known to prolong QT interval will be excluded. History of congested heart failure (CHF), or myocardial infarction (MI) or stroke in the last 3 months will be excluded.
12. Had active illicit drug use or diagnosis of alcoholism.
13. Had tumors with known IDH1 (isocitrate dehydrogenase 1) or known IDH2 mutations as determined by immunohistochemistry for the IDH1 R132H variant or by direct sequencing. IDH1/2-mutant gliomas have a markedly longer overall survival rate compared to those with IDH1/2-wildtype glioma (Parsons et al., 2008; Yan et al., 2009), indicating IDH1/2-mutant gliomas have a distinct natural history.
14. Had tumors with known 1p/19q co-deletion.
15. Had known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ melanoma, or in situ cervical cancer that has undergone potentially curative therapy.
16. Had any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures. An interval of 1 week for stereotactic brain biopsy from the start of study treatment is acceptable.
17. Had concomitant use of potent cytochrome P450 (CYP)3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting study drug administration.
18. Had concomitant use of potent CYP3A4/5 inducers, which include enzyme inducing antiepileptic drugs (EIAEDs), during the treatment phase of the study and within 2 weeks prior to starting treatment. Concurrent dexamethasone is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Mellemed, MD, Study Director — Chimerix, Inc.
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - New York University School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Arrillaga-Romany I, Gardner SL, Odia Y, Aguilera D, Allen JE, Batchelor T, Butowski N, Chen C, Cloughesy T, Cluster A, de Groot J, Dixit KS, Graber JJ, Haggiagi AM, Harrison RA, Kheradpour A, Kilburn LB, Kurz SC, Lu G, MacDonald TJ, Mehta M, Melemed AS, Nghiemphu PL, Ramage SC, Shonka N, Sumrall A, Tarapore RS, Taylor L, Umemura Y, Wen PY. ONC201 (Dordaviprone) in Recurrent H3 K27M-Mutant Diffuse Midline Glioma. J Clin Oncol. 2024 May 1;42(13):1542-1552. doi: 10.1200/JCO.23.01134. Epub 2024 Feb 9. PMID 38335473

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 43 | 30
Completed | 0 | 0
Not Completed | 43 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 43 | 30 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 29 | 69
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 38.6 [20 to 72] | 35.0 [21 to 66] | 37.1 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 33
  Male | 22 | 18 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 40 | 23 | 63
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 30 | 21 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Primary Tumor Location/Diagnosis [Count of Participants; unit: Participants]
  Brainstem (excluding DIPG) | 7 | 3 | 10
  Midline (excluding brainstem, DIPG, and spinal) | 26 | 20 | 46
  Non-midline | 1 | 7 | 8
  DIPG | 2 | 0 | 2
  Spinal | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Overall Response
Description: Quantitative thresholds for objective response by Response Assessment in Neuro-Oncology (RANO) criteria for target lesions on radiographic imaging are Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) requires a ≥50% decrease in the sum of products of perpendicular diameters of target lesions from baseline. Other considerations for RANO response include assessments of non-target lesions, corticosteroids, and performance status. The Overall Response Rate is the proportion of patients who achieve either CR or PR. Tumor assessments were conducted at 8 weeks (±1 week) following the initiation of therapy and every 8 weeks (±1 week) thereafter.
  All patients who received at least one dose of dordaviprone (ONC201) were included in the analysis, including patients with diffuse intrinsic pontine glioma (DIPG) or primary spinal tumors, which are historically not assessable for response using RANO-HGG criteria due to anatomical or imaging limitations.
Time Frame: From first dose of study treatment through study completion, an average of 1 year
Population: Note: A total of 9 (21%) patients in Arm A, including 7 with primary spinal tumors and 2 with DIPG, were included in the overall analysis (i.e. Overall Response Rate) despite not being assessable for response per RANO-HGG.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Patients received 625 mg dordaviprone (ONC201) once weekly.
  Arm A included patients with recurrent H3 K27M-mutant glioma including those with diffuse intrinsic pontine glioma (DIPG), primary spinal tumors, and some atypical histologies. Notably, patients with DIPG and primary spinal tumors are historically not evaluable for response using RANO-HGG criteria.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 43 | 30
Participants | 5 | 5

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first documented response to the earliest date of disease progression or death, whichever occurred first. Patients who had not progressed or died at the time of analysis were censored at their last adequate tumor assessment.
Time Frame: From objective response (complete response or partial response) per RANO to disease progression or death, up to 40.6 months.
Population: This outcome was analyzed in patients who achieved an objective response (complete response or partial response) per RANO criteria.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 5 | 5
months | 5.6 [1.9 to NA] — Not calculable. The statistical procedure did not have sufficient information (insufficient number of patients with events) in order to calculate the upper bound of the 95% confidence interval (CI). | 15.0 [7.5 to NA] — Not calculable. The statistical procedure did not have sufficient information (insufficient number of patients with events) in order to calculate the upper bound of the 95% confidence interval (CI).

ADVERSE EVENTS:
Time Frame: From the time/date of initiation of study treatment through 30 days following cessation of study treatment (regardless of treatment duration), or for duration of study treatment until initiation of other anticancer therapy, whichever occurred first, up to 51 months
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 33/43 | 25/30
Serious Adverse Events (participants affected / at risk) | 17/43 | 7/30
Other Adverse Events (participants affected / at risk) | 42/43 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=43) | Arm B (N=30)
Sinus tachycardia (Cardiac disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 4 | 1
Hydrocephalus (Nervous system disorders) | 4 | 0
Brain oedema (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=43) | Arm B (N=30)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 4
Diplopia (Eye disorders) | 2 | 6
Vision blurred (Eye disorders) | 3 | 2
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 13 | 5
Vomiting (Gastrointestinal disorders) | 8 | 3
Dysphagia (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 14 | 13
Gait disturbance (General disorders) | 10 | 6
Oedema peripheral (General disorders) | 2 | 5
Pyrexia (General disorders) | 2 | 3
Asthenia (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 6 | 0
COVID-19 (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 9 | 6
Alanine aminotransferase increased (Investigations) | 6 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 2
Lymphocyte count decreased (Investigations) | 8 | 0
Platelet count decreased (Investigations) | 5 | 1
Weight increased (Investigations) | 2 | 4
White blood cell count decreased (Investigations) | 3 | 3
Blood bilirubin increased (Investigations) | 4 | 0
Blood glucose increased (Investigations) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 10 | 7
Dizziness (Nervous system disorders) | 6 | 4
Hemiparesis (Nervous system disorders) | 4 | 4
Dysarthria (Nervous system disorders) | 4 | 3
Encephalopathy (Nervous system disorders) | 4 | 2
Memory impairment (Nervous system disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 3 | 3
Tremor (Nervous system disorders) | 2 | 4
Aphasia (Nervous system disorders) | 3 | 1
Hydrocephalus (Nervous system disorders) | 4 | 0
Depressed level of consciousness (Nervous system disorders) | 3 | 0
Seizure (Nervous system disorders) | 0 | 3
Confusional state (Psychiatric disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Urinary incontinence (Renal and urinary disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Hypertension (Vascular disorders) | 3 | 3
Cushingoid (Endocrine disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
The Sponsor terminated this study based on the initiation of a randomized Phase 3 study of dordaviprone (ONC201) in an earlier setting; closing this study ensured enrollment would not compete with the Phase 3 study. The decision was not related to any safety concerns with dordaviprone (ONC201). At the time enrollment was halted, some treatment arms had not completed enrollment.

Note: This study did not assess response using RANO 2.0, as these criteria were established after study initiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months of the completion of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given the opportunity to review and comment. Institution publications may be delayed up to an additional 90 days to allow the Sponsor to seek patent protection.

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03295396/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT03295396/SAP_001.pdf